CLINICAL TRIAL: NCT04690127
Title: The Effects of Plyometric Training on Vastus Lateralis and Biceps Femoris Muscle Architectures in Individuals Undergoing Anterior Cruciate Ligament Reconstruction
Brief Title: Muscle Architecture and Anterior Cruciate Ligament
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Murat EMİRZEOĞLU, Physiotherapist (MSc), Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-11167
Record Dates: First submitted 2020-12-19; First posted 2020-12-30 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: biceps femoris; vastus lateralis; muscle architecture; anterior cruciate ligament; plyometric training; action observation; motor imagery; fiber length; pennation angle; muscle thickness; function
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: Parallel group randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric Training Group (Experimental): Individuals in the plyometric training group will receive plyometric training. In this training, individuals will not participate in a real plyometric training. Volunteers will watch videos to be prepared (action observation) and imagine them performing those exercises (motor imagery). Except for one session that will be applied every two weeks, all other trainings will be given on the basis of telerehabilitation via distance education tools.
  Interventions: Other: Plyometric Exercise
- Control Group (No Intervention): Volunteers in this group will not participate in any training.

INTERVENTIONS:
Other: Plyometric Exercise — Plyometric training consisting of ten different exercises [vertical unilateral and bilateral counter movement jump, horizontal unilateral and bilateral counter movement jump, drop jump (30 cm), squat jump, step-hop (20 cm), 180 degree rotation in transverse plane, frontal plane hurdle jump (20 cm) and sagittal plane hurdle jump (20 cm)] for 8 weeks, 3 sessions per week. Individuals will not participate in a real plyometric training. Volunteers will watch videos to be prepared (action observation) and imagine them performing those exercises (motor imagery)
  Arms: Plyometric Training Group

SUMMARY:
The aim of this study is to examine the effects of plyometric training on biceps femoris longus (BFl) and vastus lateralis (VL) muscle architecture in individuals with anterior cruciate ligament reconstruction (ACLR). Individuals will be randomly placed into training and control groups. Measurements of muscle architecture will be taken bilaterally from BFl and VL muscles by means of an ultrasound device. Functional performance will be evaluated with the International Knee Documentation Committee score and the single leg jump test. Following the initial evaluations, individuals in the training group will receive plyometric training. Evaluations of muscle architecture and functional performance will be taken again from the individuals in the training and control groups at the end of the 4th and 8th weeks. The received ultrasound images will be calculated through the MicroDicom software. In-group and between-group comparisons will be analyzed using the Statistical Package for the Social Sciences program and appropriate tests.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) injuries are common, especially in young individuals participating in rolling and jumping activities. After injury, many people undergo ACL reconstruction (ACLR) surgery. The aim of this study is to examine the effects of plyometric training on biceps femoris longus (BFl) and vastus lateralis (VL) muscle architecture (fiber length, penation angle and muscle thickness) in individuals with ACLR. Individuals who have undergone ACLR in this study, which is designed as a parallel group randomized controlled study, will be randomly placed into two different groups, the training group and the control group. Imagery ability, self-efficacy and motivation will be evaluated with various questionnaires and scales in order to compare the homogeneity of the groups. Measurements of muscle architecture will be taken bilaterally from BFl and VL muscles by means of an ultrasound device. Functional performance will be evaluated with the International Knee Documentation Committee score and the single leg jump test. Following the initial evaluations, individuals in the training group will receive plyometric training consisting of ten different exercises for 8 weeks, 3 sessions per week. In this training, individuals will not participate in a real plyometric training. Volunteers will watch videos to be prepared (action observation) and imagine them performing those exercises (motor imagery). Except for one session that will be applied every two weeks, all other trainings will be given on the basis of telerehabilitation via distance education tools. Cognitive fatigue at the beginning and end of the session; at the end of each session, the technical quality and efficiency of the training will be evaluated. Evaluations of muscle architecture and functional performance will be taken again from the individuals in the control and training groups at the end of the 4th and 8th weeks. The received ultrasound images will be calculated through the MicroDicom software. In-group and between-group comparisons will be analyzed using the Statistical Package for the Social Sciences program and appropriate tests.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with unilateral anterior cruciate ligament reconstruction (ACLR)
* Volunteers using hamstring autograft in their ACLR
* Volunteers who have passed 1-5 years after their ACLR

Exclusion Criteria:

* Those who underwent same-side meniscus repair other than ACLR
* Those who have had revision surgery
* Those who had posterior cruciate ligament rupture in addition to anterior cruciate ligament
* Third-degree tears in the lateral or medial collateral ligaments
* Those with 2nd or 3rd degree strain injuries in hamstring and quadriceps muscle groups
* Those with a history of congenital, neurological, orthopedic, rheumatologic and cardiopulmonary pathology or anomalies,
* Those with serious systemic diseases

Relative Exclusion Criteria:

* Those with acute infection or pain
* Those with joint instability
* Those with a body mass index of 30 and above
* Those receiving energy supplements or ergogenic assistance during or during the 6-month period prior to work

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Muscle Architecture Change-1 | Before, at the end of the fourth week and the eighth week
  Fiber length of the vastus lateralis and biceps femoris longus muscles
Muscle Architecture Change-2 | Before, at the end of the fourth week and the eighth week
  Pennation angle of the vastus lateralis and biceps femoris longus muscles
Muscle Architecture Change-3 | Before, at the end of the fourth week and the eighth week
  Muscle thickness of the vastus lateralis and biceps femoris longus muscles

SECONDARY OUTCOMES:
Functional Performance Change-1 | Before, at the end of the fourth week and the eighth week
  International knee documentation committee score. (Minimum score: 0 Maximum score: 100. Higher scores mean a better outcome.
Functional Performance Change-2 | Before, at the end of the fourth week and the eighth week
  Single leg jump distance

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe Üniversitesi, Ankara, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No